CLINICAL TRIAL: NCT02274701
Title: Evaluating the Impact of Holistic Needs Assessment in Outpatient Cancer Care
Brief Title: Holistic Needs Assessment in Outpatient Cancer Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of the West of Scotland (Other)
Collaborators: Macmillan Cancer Support (Other)
Responsible Party: Principal Investigator, Jenny Young, Mrs Jenny Young, University of the West of Scotland
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: 14/WS/0126
Record Dates: First submitted 2014-10-16; First posted 2014-10-24 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Oncology [See Also, Affected System]

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Holistic Needs Assessment (Experimental): Participants (patients) complete a self-reported paper assessment that asks them to indicate whether they have any emotional, practical, financial and/or clinical concerns. The patient then takes this completed assessment into their consultation. It is then given to the clinician where it informs a discussion based on the patient's needs and concerns as identified by them. A care plan is then written based on this assessment.
  Interventions: Other: Holistic Needs Assessment
- Control (No Intervention): The control group entails standard care - routine consultation between the patient and clinician.

INTERVENTIONS:
Other: Holistic Needs Assessment — An assessment completed by the patient in cancer care. It is recommended that this assessment is completed at key points in the care pathway, such as at diagnosis, post treatment and beginning of end of life care. The aim of this assessment is to allow the patient to discuss their most important needs as identified by them. The clinician will take any appropriate action. This may range from listening to the patient to referring to another member of the multi-disciplinary team.
  Other Names: The Concerns Checklist
  Arms: Holistic Needs Assessment

SUMMARY:
This study evaluates the impact of holistic needs assessment (HNA) on patient/clinician communication in outpatient cancer care. Half of the participants will complete a HNA prior to their clinical consultation. They will then take it into the consultation and it will inform a discussion around any identified areas of need. Half of the participants will be in the control group meaning there will be no additional intervention they will receive care as normal. The consultations will be audio-recorded. The patient will complete two outcome measures following the consultation.

DETAILED DESCRIPTION:
Holistic needs assessment is a checklist completed by the patient prior to consultation. It signposts issues of emotional, practical, financial and clinical concern. The purpose of a HNA is to identify patient's individual needs in order to facilitate better collaboration. During consultation the HNA facilitates a dialogue that will have the patient's concerns at the centre. In conjunction with a subsequent care plan the process supports timely intervention based on a collaborative, person centred discussion. However, there is little evidence on how HNA impacts upon the dynamics of the clinical consultation. This study aims to establish a) how HNA affects the type of conversation that goes on during a clinical consultation and b) how these putative changes impact on shared decision-making and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18, capable of informed consent and expresses a wish to participate.
* Diagnosed with cancer and attending a post-treatment out-patient oncology clinic.

Exclusion Criteria:

* Individuals not diagnosed with cancer.
* Non English speaker
* Person deemed incapable of consenting to participate as defined by the Adults with Incapacity Act (2000)
* Any reason which in the opinion of the clinician/investigator interferes with the ability of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Patient participation | This outcome measure will be collected during the patients first clinic appointment after treatment for their cancer. The consultation will last approximately 15 minutes.
  Measured through analysis of the audio-recordings from each recorded consultation between a clinician and patient. Specifically, through measuring dialogue ratio and preponderance of initiative. These two measures indicate who is speaking, when and for how long.

SECONDARY OUTCOMES:
Shared decision making | This outcome measure will be collected following the patients first clinic appointment after treatment. The patient will return to the researcher and complete this measure. It is expected to take no more than 1 minute to complete.
  Measured through patient self-report using the measure CollaboRATE. CollaboRATE is a survey-based validated tool designed to create a fast way to measure how much effort clinicians make to explain their patients' health issues; how much effort they make to listen to the issues that matter most to their patients and how much effort they make to integrate the patients' views and health beliefs.
Self-efficacy | This outcome measure will be collected following the patients first clinic appointment after treatment. The patient will return to the researcher and complete this measure. It is expected to take no more than 5 minutes..
  Measured through self-report using The Lorig Self-Efficacy for Managing Chronic Disease 6-Item Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Austyn Snowden, PhD, Principal Investigator — University of the West of Scotland

REFERENCES:
- [Background] Snowden A, White CA, Christie Z, Murray E, McGowan C, Scott R. Helping the clinician help me: towards listening in cancer care. Br J Nurs. 2012 May 24-Jun 13;21(10):S18, S20-6. doi: 10.12968/bjon.2012.21.Sup10.S18. PMID 22875264
- [Background] Snowden A, White CA, Christie Z, Murray E, McGowan C, Scott R. The clinical utility of the distress thermometer: a review. Br J Nurs. 2011 Feb 24-Mar 9;20(4):220-7. doi: 10.12968/bjon.2011.20.4.220. PMID 21471860
- [Derived] Snowden A, Young J, Roberge D, Schipani S, Murray E, Richard C, Lussier MT, White C. Holistic needs assessment in outpatient cancer care: a randomised controlled trial. BMJ Open. 2023 May 4;13(5):e066829. doi: 10.1136/bmjopen-2022-066829. PMID 37142317
- [Derived] Snowden A, Young J, White C, Murray E, Richard C, Lussier MT, MacArthur E, Storey D, Schipani S, Wheatley D, McMahon J, Ross E. Evaluating holistic needs assessment in outpatient cancer care--a randomised controlled trial: the study protocol. BMJ Open. 2015 May 11;5(5):e006840. doi: 10.1136/bmjopen-2014-006840. PMID 25967990